CLINICAL TRIAL: NCT06315088
Title: BIOQUALIM: From Cultivated Biodiversity to Prevention in Human Health
Brief Title: Food Biodiversity and Human Health
Acronym: BIOQUALIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL24_0144
Record Dates: First submitted 2024-03-01; First posted 2024-03-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Oral Microbiota; Periodontal Diseases
Keywords: biodiversity; diet; environmental and medical impact; oral health; oral microbiota; general health; quality of life
MeSH Terms: conditions — Periodontal Diseases | interventions — Health Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Einkorn Diet (Experimental): Healthy adult volunteers (not suffering from chronic pathologies) and non-smokers, having an omnivorous diet, and agreeing to change their eating habits for 3 months (reducing meat consumption by half and replacing it with einkorn).
  Interventions: Other: Einkorn Diet; Other: Intermediate oral microbiota; Other: Periodontal health status; Other: General health status

INTERVENTIONS:
Other: Einkorn Diet — Analysis of the oral microbiota before (T0) and after (T2) introduction of einkorn into the diet by interdental sampling, on 4 sites, pooled then analyzed by bacterial PCR.
  Other Names: Total Oral microbiota
Other: Intermediate oral microbiota — Comparison of the number of total bacteria and pathogens of the interdental microbiota before (T0) and in interim analysis (T1) for evaluation of the minimum period of effectiveness, by interdental sampling, on 4 sites, pooled then analyzed by bacterial PCR.
Other: Periodontal health status — Analysis of the periodontal and oral clinical parameters (plaque index, gingival index, interdental inflammation, pocket depth and loss of clinical attachment, salivary pH) before (T0) and after (T2) introduction of einkorn into the diet, by sampling and periodontal analysis of all of the participants' teeth
Other: General health status — Analysis of general health indicators (body mass index, measurement of abdominal circumference, blood pressure, MOS SF-36 quality of life questionnaire and eating habits) before (T0) and after (T2) introduction of einkorn in the diet

SUMMARY:
In Western countries, one of the major nutritional challenges requires reducing the proportion of animal proteins and increasing the proportion of vegetable proteins in the daily plate. Added to this nutritional challenge is an environmental challenge, with plant proteins being much less expensive to produce. However, plant proteins are mainly provided by cereals and legumes, a large diversity of which is necessary to cover the recommended daily intake of amino acids. However, given the collapse of cultivated biodiversity (loss of 75% in 100 years, FAO), the diversity of the supply is very reduced.

Furthermore, for several years, public health studies have indicated a chronic deficit in micronutrients (minerals/trace elements, vitamins, antioxidants) as well as fiber in the diet of the French population. This comes in particular from the impoverishment of the nutritional quality of the fruits/vegetables/cereals/legumes consumed. In general, diet plays a major role in the primary prevention of chronic diseases (cardiovascular, diabetes, cancer) including periodontal disease. Thus, a diet low in sugars, saturated fats and rich in fiber would reduce the appearance of periodontal disease by strengthening salivary capacity. However, certain pathogenic periodontal bacteria (such as Porphyromonas gingivalis) can migrate (blood, digestive or respiratory routes) to reach other organs and represent a risk factor for other chronic diseases. Thus, the prevention of periodontal diseases through diet control would also contribute to the prevention of other chronic diseases.

The benefit of plant-based diets to reduce the risk of cancer is now established. In addition, certain cereals such as spelled have superior nutritional qualities to common wheat, notably their protein content and they also contain higher quantities of certain bioactive compounds with anti-cancer properties (such as phytosterols).

Furthermore, the potential impact of the oral microbiota on chronic diseases is now being studied: in healthy adults, a dysbiotic periodontal microbiota may be likely to lead to systemic para-inflammation. It has also been shown that a dietary change (Mediterranean diet) could lead to a reduction in pathogenic bacteria in the oral microbiota (including P. gingivalis). However, the link between the introduction of cereals into the diet and the evolution of cancer risk factor bacteria in the oral microbiota has never been demonstrated.

This pilot clinical study plans to focus on the oral microbiota, with the aim of objectivizing a possible link between a modification of the diet by the introduction of cereals (einkorn type) and the evolution of certain bacteria of this microbiota. , notably P. gingivalis (but also T. forsythia, S. anginosus, A. actinomycetemcomitans, T. denticola and F. nucleatum), considered as cancer risk factors and thus observe an improvement in health status oral and general.

ELIGIBILITY:
Inclusion Criteria:

* Person between 20 and 60 years old
* Person with an omnivorous diet
* Person who has given free, informed, express written consent
* Person affiliated to a French social security system
* Person with a body mass greater than 18 kg/m²
* Person able to attend at least 1 culinary workshop

Exclusion Criteria:

* Person with a smoking addiction
* Person with a known food allergy/intolerance
* Person unable to consume dairy or solid products (e.g. chocolate milk pudding, chocolate jelly)
* Person participating in another study related to nutrition
* Patients at high risk of infective endocarditis
* Person with chronic pathologies
* Person having taken antibiotic treatment during the month preceding the start of the study
* Pregnant, parturient or breastfeeding woman
* Minors
* Persons deprived of liberty by a judicial or administrative decision
* People receiving psychiatric care
* Persons admitted to a health or social establishment for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Person with fewer than 20 natural teeth
* Person performing interdental hygiene and/or daily mouthwashes.
* Person wearing orthodontic appliance
* Person with periodontal disease (stage ≥ II periodontal lesions according to the Chicago 2017 classification (i.e. PD ≥ 4 mm, and/or CAL ≥ 4 mm) and/or generalized (>30% of sites )), active caries or during dental care

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Total periodontal bacteria count | Baseline (T0), 3 months after baseline (T2)
  Comparison of the number of total bacteria and pathogens of the interdental microbiota before (T0) and after (T2) introduction of einkorn into the diet, by interdental sampling, on 4 sites, pooled then analyzed by bacterial PCR.

SECONDARY OUTCOMES:
Intermediate periodontal bacteria count | Baseline (T0), 1 month later (T1)
  Comparison of the number of total bacteria and pathogens of the interdental microbiota before (T0) and in interim analysis (T1) for evaluation of the minimum period of effectiveness, by interdental sampling, on 4 sites, pooled then analyzed by bacterial PCR.
Periodontal health analysis:plaque index | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of periodontal and oral clinical parameters (plaque index) before (T0), intermediate (T1) and after (T2) introduction of einkorn into the diet, by sampling and periodontal analysis of all of the participants' teeth
Periodontal health analysis: gingival index | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of periodontal and oral clinical parameters (gingival index) before (T0), intermediate (T1) and after (T2) introduction of einkorn into the diet, by sampling and periodontal analysis of all of the participants' teeth
Periodontal health analysis : pocket depth and loss of clinical attachment | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of periodontal and oral clinical parameters (pocket depth and loss of clinical attachment) before (T0), intermediate (T1) and after (T2) introduction of einkorn into the diet, by sampling and periodontal analysis of all of the participants' teeth
Periodontal health analysis : interdental inflammation | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of periodontal and oral clinical parameters (interdental inflammation) before (T0), intermediate (T1) and after (T2) introduction of einkorn into the diet, by sampling and periodontal analysis of all of the participants' teeth
Periodontal health analysis : salivary pH | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of periodontal and oral clinical parameters (salivary pH) before (T0), intermediate (T1) and after (T2) introduction of einkorn into the diet, by sampling and periodontal analysis of all of the participants' teeth
General health analysis : body mass index | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of general health indicators (body mass index) before (T0), intermediate (T1) and after (T2) introduction of einkorn in the diet, by a consultation and a general medical examination
General health analysis : measurement of abdominal circumference | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of general health indicators (measurement of abdominal circumference) before (T0), intermediate (T1) and after (T2) introduction of einkorn in the diet, by a consultation and a general medical examination
General health analysis : blood pressure | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of general health indicators (blood pressure) before (T0), intermediate (T1) and after (T2) introduction of einkorn in the diet, by a consultation and a general medical examination
General health analysis : MOS SF-36 quality of life questionnaire | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of general health indicators (MOS SF-36 quality of life questionnaire) before (T0), intermediate (T1) and after (T2) introduction of einkorn in the diet, by a consultation and a general medical examination
General health analysis : eating habits | Baseline (T0), 1 month later (T1), 3 months after baseline (T2)
  Comparison of general health indicators (eating habits) before (T0), intermediate (T1) and after (T2) introduction of einkorn in the diet, by a consultation and a general medical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Maison des professionnels, Lyon, France